CLINICAL TRIAL: NCT03198000
Title: A Single-Center, Randomized, Controlled Study to Evaluate the Efficacy of Two Investigational OTC Eye Drops in Healthy Adults With Red Eye
Brief Title: A Study to Evaluate the Efficacy of Investigational OTC Eye Drops
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Consumer Inc. (J&JCI) (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CO-161103095739-VCCT
Record Dates: First submitted 2017-06-22; First posted 2017-06-23 (Actual); Results first posted 2018-08-08 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-04

CONDITIONS: Ophthalmic Solutions
Keywords: Eye Redness; Eye Comfort; Red Eyes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Formula # 13418-148 (Experimental)
  Interventions: Drug: F# 13418-148 Eye Drops
- Formula # 13418-158 (Experimental)
  Interventions: Drug: F#13418-158 Eye Drops
- Control Formula # PF004390 (Active Comparator)
  Interventions: Drug: F# PF-004390 Eye Drops

INTERVENTIONS:
Drug: F# 13418-148 Eye Drops — ocular clear liquid. Tetrahydrozoline 0.05%; Glycerin 0.40% 1-2 drops will be instilled as instructed over one day
  Arms: Formula # 13418-148
Drug: F#13418-158 Eye Drops — ocular clear liquid Tetrahydrozoline 0.05%; Glycerin 0.20%, Hypromellose 0.2%, Polyethylene glycol 400 1.0% 1-2 drops will be instilled as instructed over one day
  Arms: Formula # 13418-158
Drug: F# PF-004390 Eye Drops — Ocular clear liquid Tetrahydrozoline 0.05%; 1-2 drops will be instilled as instructed over one day
  Arms: Control Formula # PF004390

SUMMARY:
This is a single center, double-blinded study designed to demonstrate the therapeutic equivalence of over-the-counter eye drops in healthy adults with red eyes.

DETAILED DESCRIPTION:
Eligible participants will use assigned eye drop products as directed. Participants will be required to attend 2 consecutive clinic visits. Assessments for eye redness and eye comfort will be completed. Participants will complete brief questionnaires about their eyes.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to comprehend and follow the requirements of the study (including availability on scheduled visit dates) based upon research site personnel's assessment;
2. Able and willing to provide a signed and dated Informed Consent document and Authorization for the Release of Health Information for Research
3. Male or female of any race or ethnicity, aged 18 years and older;
4. Females of childbearing potential who have a negative urine pregnancy test at the Screening/Baseline visit (Visit 1);
5. Able to read and understand English;
6. Healthy subjects with redness in both eyes
7. History of topical ocular drugs or desire to use within the last 6 months;
8. Ocular health within normal limits,
9. Male and female subjects with reproductive potential who agree to practice a medically acceptable form of birth control during the study and for 30 days following the last dose of investigational product. Females must have used such birth control for at least 3 months prior to the Screening/Baseline Visit 1.

Exclusion Criteria:

1. Suspected alcohol or substance abuse (e.g., amphetamines, benzodiazepines, cocaine, marijuana, opiates);
2. Known sensitivity, allergy or contraindications to any investigational product ingredient;
3. Females who are pregnant, planning to become pregnant or breastfeeding during the study;
4. Subjects who were previously screened and determined to be ineligible for the study;
5. Use of a therapeutic eye treatment (over-the-counter or prescription) within 2 days of the Screening/Baseline visit (Visit 1) and throughout study participation;
6. Participation in any clinical study investigation within 30 days of Screening/Baseline visit (Visit 1);
7. Relative, partner or staff of any clinical research site personnel;
8. Active infection of any type at the start of the study; particularly, presence of active ocular infection (bacterial, viral, or fungal) or positive history of an ocular herpetic infection;
9. Any ocular condition that could affect the subject's safety or trial parameter, such as severe ocular allergy;
10. Planned surgery during the trial period, 6 months prior to clinic visit 1 or 30 days after the end of study period;
11. Has a compromised immune system;
12. Has any acute or chronic, medical or psychiatric conditions
13. Contact lens use within 24 hours prior to clinic Visit 1 and during their participation in the study;
14. Saline eye drop use within 24 hours prior to clinic Visit 1 and during their participation in the study;
15. Use of any new OTC or prescription medications within 24 hours prior to clinic Visit 1 and throughout study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2017-06-28 (Actual); Primary Completion 2017-07-21 (Actual); Study Completion 2017-07-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail Torkildsen, MD, Principal Investigator — Andover Eye Associates
Locations (1):
- Andover Eye Associates, Andover, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cronau H, Kankanala RR, Mauger T. Diagnosis and management of red eye in primary care. Am Fam Physician. 2010 Jan 15;81(2):137-44. PMID 20082509
- [Background] Hara JH. The red eye: diagnosis and treatment. Am Fam Physician. 1996 Dec;54(8):2423-30. PMID 8961843
- [Background] Murphy PJ, Lau JS, Sim MM, Woods RL. How red is a white eye? Clinical grading of normal conjunctival hyperaemia. Eye (Lond). 2007 May;21(5):633-8. doi: 10.1038/sj.eye.6702295. Epub 2006 Mar 3. PMID 16518366

RESULTS

PARTICIPANT FLOW:
Groups:
- F#13418-148/F#13418-158: Eye drops - one formula in each eye: Formula #13418-148 = tetrahydrozoline 0.05%, glycerin 0.40%; Formula #13418-158 = tetrahydrozoline 0.05%, glycerin 0.20%, hypromellose 0.20%, polyethylene glycol 400 1.0%
- F#13418-148/F#PF004390: Eye drops - one formula in each eye: Formula #13418-148 = tetrahydrozoline 0.05%, glycerin 0.40%; Formula #PF004390 = tetrahydrozoline 0.05%
- F#13418-158/F#PF004390: Eye drops - one formula in each eye: Formula #13418-158 = tetrahydrozoline 0.05%, glycerin 0.20%, hypromellose 0.20%, polyethylene glycol 400 1.0%; Formula #PF004390 = tetrahydrozoline 0.05%
Period: Overall Study
Arm/Group | F#13418-148/F#13418-158 | F#13418-148/F#PF004390 | F#13418-158/F#PF004390
Started | 41 | 38 | 41
Completed | 41 | 38 | 41
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | F#13418-148/F#13418-158 | F#13418-148/F#PF004390 | F#13418-158/F#PF004390 | Total
Number analyzed (Participants) | 41 | 38 | 41 | 120
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Intent-to-treat set
  Years | 55.4 (15.58) | 59.1 (13.85) | 54.9 (12.47) | 56.4 (14.03)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Intent-to-treat set
  Participants
    Female | 27 | 22 | 26 | 75
    Male | 14 | 16 | 15 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Intent-to-treat set
  Participants
    White | 36 | 36 | 39 | 111
    Black or African-American | 3 | 1 | 0 | 4
    Asian | 1 | 0 | 1 | 2
    Other | 1 | 1 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Intent-to-treat set
  Participants
    Hispanic or Latino | 1 | 3 | 7 | 11
    Not Hispanic or Latino | 40 | 35 | 34 | 109
Region of Enrollment [Count of Participants; unit: Participants] — Population: Intent-to-treat set
  Participants
    United States | 41 | 38 | 41 | 120

OUTCOME MEASURES:

1. Primary Outcome: Clinician Assessment of Change From Baseline in Redness at 60 Seconds After First Product Application
Description: Mean change from baseline in redness. Redness was assessed on a 5-point severity scale with 0.5 increments (0 = none, 1 = mild, 2 = moderate, 3 = severe, and 4 = extremely severe), where a lower score is better.
Time Frame: Baseline to 60 seconds after first product application
Population: Intent-to-treat set
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: eyes
Groups:
- F# PF004390 Eye Drops: Active Comparator - Tetrahydrozoline 0.05%
- F# 13418-148 Eye Drops: Experimental - Tetrahydrozoline 0.05%; glycerin 0.40%
- F#13418-158 Eye Drops: Experimental - Tetrahydrozoline 0.05%; glycerin 0.20%; hypromellose 0.20%; polyethylene glycol 400 1.0%
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (eyes) | 79 | 79 | 82
units on a scale | 0.31 (0.050) | 0.27 (0.050) | 0.32 (0.049)
Statistical Analysis 1: Comparison: F# PF004390 Eye Drops vs F# 13418-148 Eye Drops; Test type: Equivalence — Prespecified equivalence interval of (-0.22, 0.44); p = 0.392, ANCOVA; Mixed effect ANCOVA with treatment as factor and baseline value as a covariate; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.140 to 0.055], Standard Error of Mean 0.049
Statistical Analysis 2: Comparison: F# PF004390 Eye Drops vs F#13418-158 Eye Drops; Test type: Equivalence — Prespecified equivalence interval of (-0.22, 0.44); p = 0.828, ANCOVA; Mixed effect ANCOVA with treatment as factor and baseline value as a covariate; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.086 to 0.107], Standard Error of Mean 0.049

2. Primary Outcome: Percentage of Participants With Response to Redness at 60 Seconds After First Product Application
Description: The responder was defined as a subject whose assessment score at 60 seconds after the initial eye drop is less than the assessment score at baseline. Redness was assessed on a 5-point severity scale with 0.5 increments (0 = none, 1 = mild, 2 = moderate, 3 = severe, and 4 = extremely severe), where a lower score is better.
Time Frame: Baseline to 60 seconds after first product application
Population: Intent-to-treat set
Measure: Number; unit: Percentage
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage | 53.6 | 50.1 | 50.1
Statistical Analysis 1: Comparison: F# PF004390 Eye Drops vs F# 13418-148 Eye Drops; Test type: Equivalence — Prespecified equivalence interval of (0.80, 1.25); p = 0.576, GEE model; GEE model with treatment as factor; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.539 to 1.411]
Statistical Analysis 2: Comparison: F# PF004390 Eye Drops vs F#13418-158 Eye Drops; Test type: Equivalence — Prespecified equivalence interval of (0.80, 1.25); p = 0.544, GEE model; GEE model with treatment as factor; Odds Ratio (OR) = 0.87, 95% CI 2-sided [0.552 to 1.368]

3. Secondary Outcome: Clinician Assessment of Change From Baseline in Redness at 30 Seconds After First Product Application
Description: as for outcome 1
Time Frame: Baseline to 30 seconds after first product application
Population: Intent-to-treat set
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (eyes) | 79 | 79 | 82
units on a scale | 0.10 (0.046) | 0.09 (0.046) | 0.11 (0.046)
Statistical Analysis 1: Comparison: F# PF004390 Eye Drops vs F# 13418-148 Eye Drops; Test type: Equivalence — No equivalence interval was specified for this time point; p = 0.893, ANCOVA; Mixed effect ANCOVA with treatment as factor and baseline value as a covariate; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.085 to 0.074], Standard Error of Mean 0.040
Statistical Analysis 2: Comparison: F# PF004390 Eye Drops vs F#13418-158 Eye Drops; Test type: Equivalence — No equivalence interval was specified for this time point; p = 0.886, ANCOVA; Mixed effect ANCOVA with treatment as factor and baseline value as a covariate; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.073 to 0.084], Standard Error of Mean 0.040

4. Secondary Outcome: Clinician Assessment of Change From Baseline in Redness at 2 Minutes After First Product Application
Description: as for outcome 1
Time Frame: Baseline to 2 minutes after first product application
Population: Intent-to-treat set
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (eyes) | 79 | 79 | 82
units on a scale | 0.88 (0.048) | 0.80 (0.048) | 0.83 (0.048)
Statistical Analysis 1: Comparison: F# PF004390 Eye Drops vs F# 13418-148 Eye Drops; Test type: Equivalence — No equivalence interval was specified for this time point; p = 0.117, ANCOVA; Mixed effect ANCOVA with treatment as factor and baseline value as a covariate; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.177 to 0.020], Standard Error of Mean 0.050
Statistical Analysis 2: Comparison: F# PF004390 Eye Drops vs F#13418-158 Eye Drops; Test type: Equivalence — No equivalence interval was specified for this time point; p = 0.255, ANCOVA; Mixed effect ANCOVA with treatment as factor and baseline value as a covariate; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.153 to 0.041], Standard Error of Mean 0.049

5. Secondary Outcome: Clinician Assessment of Baseline Redness
Description: Redness was assessed on a 5-point severity scale with 0.5 increments (0 = none, 1 = mild, 2 = moderate, 3 = severe, and 4 = extremely severe), where a lower score is better.
Time Frame: Baseline
Population: Intent-to-treat set
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (eyes) | 79 | 79 | 82
units on a scale | 1.64 (0.537) | 1.66 (0.497) | 1.76 (0.498)

6. Secondary Outcome: Change From Baseline in Ocular Comfort at 60 Seconds After First Product Application
Description: Ocular comfort was assessed on an 11-point visual analog scale (0-10) where 0 = very uncomfortable and 10 = very comfortable, where a higher score was better.
Time Frame: Baseline to 60 seconds after first product application
Population: Intent-to-treat set
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (eyes) | 79 | 79 | 82
units on a scale | -1.4 (0.21) | -1.1 (0.21) | -1.2 (0.20)
Statistical Analysis 1: Comparison: F# PF004390 Eye Drops vs F# 13418-148 Eye Drops; Test type: Equivalence — No equivalence interval was specified; p = 0.085, ANCOVA; Mixed effect ANCOVA with treatment as factor and baseline value as a covariate; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.05 to 0.78], Standard Error of Mean 0.21
Statistical Analysis 2: Comparison: F# PF004390 Eye Drops vs F#13418-158 Eye Drops; Test type: Equivalence — No equivalence interval was specified for this time point; p = 0.269, ANCOVA; Mixed effect ANCOVA with treatment as factor and baseline value as a covariate; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.18 to 0.64], Standard Error of Mean 0.21

7. Secondary Outcome: Change From Baseline in Ocular Comfort at 10 Hours After First Product Application
Description: as for outcome 6
Time Frame: Baseline to 10 hours after first product application
Population: Intent-to-treat set
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (eyes) | 79 | 79 | 82
units on a scale | -1.4 (0.20) | -1.7 (0.20) | -1.6 (0.20)
Statistical Analysis 1: Comparison: F# PF004390 Eye Drops vs F# 13418-148 Eye Drops; Test type: Equivalence — No equivalence interval was specified; p = 0.162, ANCOVA; Mixed effect ANCOVA with treatment as factor and baseline value as a covariate; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.60 to 0.10], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: F# PF004390 Eye Drops vs F#13418-158 Eye Drops; Test type: Equivalence — No equivalence interval was specified for this time point; p = 0.234, ANCOVA; Mixed effect ANCOVA with treatment as factor and baseline value as a covariate; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.55 to 0.14], Standard Error of Mean 0.17

8. Secondary Outcome: Change From Baseline in Ocular Comfort at 12 Hours After First Product Application
Description: as for outcome 6
Time Frame: Baseline to 12 hours after first product application
Population: Intent-to-treat set
Measure: Mean (Standard Error); unit: units on a scale
Units Other Than Participants: eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (eyes) | 79 | 79 | 82
units on a scale | -1.4 (0.20) | -1.5 (0.20) | -1.6 (0.20)
Statistical Analysis 1: Comparison: F# PF004390 Eye Drops vs F# 13418-148 Eye Drops; Test type: Equivalence — No equivalence interval was specified; p = 0.398, ANCOVA; Mixed effect ANCOVA with treatment as factor and baseline value as a covariate; Mean Difference (Final Values) = -0.1, 95% CI 2-sided [-0.48 to 0.19], Standard Error of Mean 0.17
Statistical Analysis 2: Comparison: F# PF004390 Eye Drops vs F#13418-158 Eye Drops; Test type: Equivalence — No equivalence interval was specified for this time point; p = 0.233, ANCOVA; Mixed effect ANCOVA with treatment as factor and baseline value as a covariate; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.54 to 0.13], Standard Error of Mean 0.17

9. Secondary Outcome: My Eye Feels Hydrated - Baseline
Description: Subject questionnaire. Assessed on a 5-point scale (1-5) where 1 = strongly disagree, 2 = somewhat disagree, 3 = neither agree or disagree, 4 = somewhat agree, and 5 = strongly agree, where a higher score was better. No opinion was also allowed.
Time Frame: Baseline
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 8.9 | 10.1 | 8.5
  Somewhat agree (4) | 30.4 | 34.2 | 28.0
  Neither agree or disagree (3) | 10.1 | 12.7 | 9.8
  Somewhat disagree (2) | 30.4 | 30.4 | 34.1
  Strongly disagree (1) | 17.7 | 10.1 | 19.5
  No opinion | 2.5 | 2.5 | 0

10. Secondary Outcome: My Eye Feels Hydrated - 2 Minutes After First Application
Description: as for outcome 9
Time Frame: 2 minutes after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 45.6 | 39.2 | 43.9
  Somewhat agree (4) | 48.1 | 49.4 | 42.7
  Neither agree or disagree (3) | 3.8 | 3.8 | 7.3
  Somewhat disagree (2) | 1.3 | 6.3 | 6.1
  Strongly disagree (1) | 1.3 | 1.3 | 0
  No opinion | 0 | 0 | 0

11. Secondary Outcome: My Eye Feels Hydrated - 10 Hours After First Application
Description: as for outcome 9
Time Frame: 10 hours after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 31.6 | 43.0 | 29.3
  Somewhat agree (4) | 41.8 | 35.4 | 41.5
  Neither agree or disagree (3) | 10.1 | 8.9 | 11.0
  Somewhat disagree (2) | 11.4 | 8.9 | 13.4
  Strongly disagree (1) | 2.5 | 2.5 | 4.9
  No opinion | 1.3 | 1.3 | 0

12. Secondary Outcome: My Eye Feels Hydrated - 12 Hours After First Application
Description: as for outcome 9
Time Frame: 12 hours after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 36.7 | 35.4 | 30.5
  Somewhat agree (4) | 43.0 | 40.5 | 41.5
  Neither agree or disagree (3) | 3.8 | 6.3 | 7.3
  Somewhat disagree (2) | 12.7 | 8.9 | 17.1
  Strongly disagree (1) | 2.5 | 6.3 | 3.7
  No opinion | 0 | 0 | 0

13. Secondary Outcome: My Eye Feels Refreshed - 2 Minutes After First Application
Description: as for outcome 9
Time Frame: 2 minutes after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 38.0 | 36.7 | 42.7
  Somewhat agree (4) | 46.8 | 44.3 | 36.6
  Neither agree or disagree (3) | 7.6 | 10.1 | 14.6
  Somewhat disagree (2) | 6.3 | 8.9 | 4.9
  Strongly disagree (1) | 1.3 | 0 | 1.2
  No opinion | 0 | 0 | 0

14. Secondary Outcome: My Eye Feels Refreshed - 10 Hours After First Application
Description: as for outcome 9
Time Frame: 10 hours after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 32.9 | 34.2 | 32.9
  Somewhat agree (4) | 36.7 | 45.6 | 43.9
  Neither agree or disagree (3) | 13.9 | 3.8 | 6.1
  Somewhat disagree (2) | 13.9 | 15.2 | 9.8
  Strongly disagree (1) | 1.3 | 1.3 | 7.3
  No opinion | 0 | 0 | 0

15. Secondary Outcome: My Eye Feels Refreshed - 12 Hours After First Application
Description: as for outcome 9
Time Frame: 12 hours after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 27.8 | 30.4 | 26.8
  Somewhat agree (4) | 38.0 | 36.7 | 37.8
  Neither agree or disagree (3) | 16.5 | 12.7 | 14.6
  Somewhat disagree (2) | 11.4 | 12.7 | 12.2
  Strongly disagree (1) | 3.8 | 5.1 | 8.5
  No opinion | 0 | 1.3 | 0

16. Secondary Outcome: The Appearance of my Eye Gives me Confidence to Approach Others - Baseline
Description: as for outcome 9
Time Frame: Baseline
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 43.0 | 30.4 | 30.5
  Somewhat agree (4) | 25.3 | 31.6 | 26.8
  Neither agree or disagree (3) | 20.3 | 20.3 | 23.2
  Somewhat disagree (2) | 1.3 | 5.1 | 8.5
  Strongly disagree (1) | 2.5 | 3.8 | 7.3
  No opinion | 7.6 | 8.9 | 3.7

17. Secondary Outcome: The Appearance of my Eye Gives me Confidence to Approach Others - 2 Minutes After First Application
Description: as for outcome 9
Time Frame: 2 minutes after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 46.8 | 39.2 | 37.8
  Somewhat agree (4) | 24.1 | 32.9 | 36.6
  Neither agree or disagree (3) | 20.3 | 11.4 | 15.9
  Somewhat disagree (2) | 1.3 | 3.8 | 2.4
  Strongly disagree (1) | 1.3 | 2.5 | 4.9
  No opinion | 6.3 | 10.1 | 2.4

18. Secondary Outcome: The Appearance of my Eye Gives me Confidence to Approach Others - 10 Hours After First Application
Description: as for outcome 9
Time Frame: 10 hours after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 46.8 | 51.9 | 46.3
  Somewhat agree (4) | 29.1 | 26.6 | 28.0
  Neither agree or disagree (3) | 10.1 | 8.9 | 14.6
  Somewhat disagree (2) | 6.3 | 6.3 | 4.9
  Strongly disagree (1) | 0 | 1.3 | 2.4
  No opinion | 6.3 | 5.1 | 3.7

19. Secondary Outcome: The Appearance of my Eye Gives me Confidence to Approach Others - 12 Hours After First Application
Description: as for outcome 9
Time Frame: 12 hours after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 38.0 | 38.0 | 30.5
  Somewhat agree (4) | 36.7 | 32.9 | 37.8
  Neither agree or disagree (3) | 15.2 | 13.9 | 18.3
  Somewhat disagree (2) | 1.3 | 1.3 | 3.7
  Strongly disagree (1) | 0 | 5.1 | 3.7
  No opinion | 7.6 | 7.6 | 6.1

20. Secondary Outcome: The Appearance of my Eye Can Show How I Really Feel - Baseline
Description: as for outcome 9
Time Frame: Baseline
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 34.2 | 29.1 | 25.6
  Somewhat agree (4) | 36.7 | 40.5 | 37.8
  Neither agree or disagree (3) | 15.2 | 16.5 | 18.3
  Somewhat disagree (2) | 3.8 | 2.5 | 9.8
  Strongly disagree (1) | 1.3 | 3.8 | 3.7
  No opinion | 8.9 | 7.6 | 4.9

21. Secondary Outcome: The Appearance of my Eye Can Show How I Really Feel - 2 Minutes After First Application
Description: as for outcome 9
Time Frame: 2 minutes after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 36.7 | 34.2 | 35.4
  Somewhat agree (4) | 34.2 | 43.0 | 40.2
  Neither agree or disagree (3) | 19.0 | 12.7 | 14.6
  Somewhat disagree (2) | 3.8 | 6.3 | 2.4
  Strongly disagree (1) | 1.3 | 0 | 2.4
  No opinion | 5.1 | 3.8 | 4.9

22. Secondary Outcome: The Appearance of my Eye Can Show How I Really Feel - 10 Hours After First Application
Description: as for outcome 9
Time Frame: 10 hours after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 35.4 | 31.6 | 32.9
  Somewhat agree (4) | 31.6 | 36.7 | 31.7
  Neither agree or disagree (3) | 20.3 | 22.8 | 24.4
  Somewhat disagree (2) | 2.5 | 2.5 | 1.2
  Strongly disagree (1) | 0 | 1.3 | 2.4
  No opinion | 8.9 | 5.1 | 7.3

23. Secondary Outcome: The Appearance of my Eye Can Show How I Really Feel - 12 Hours After First Application
Description: as for outcome 9
Time Frame: 12 hours after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 34.2 | 35.4 | 32.9
  Somewhat agree (4) | 38.0 | 36.7 | 40.2
  Neither agree or disagree (3) | 17.7 | 15.2 | 18.3
  Somewhat disagree (2) | 3.8 | 2.5 | 3.7
  Strongly disagree (1) | 0 | 1.3 | 1.2
  No opinion | 5.1 | 6.3 | 3.7

24. Secondary Outcome: My Eye Appears Healthy - Baseline
Description: as for outcome 9
Time Frame: Baseline
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 40.5 | 41.8 | 45.1
  Somewhat agree (4) | 35.4 | 31.6 | 25.6
  Neither agree or disagree (3) | 10.1 | 15.2 | 8.5
  Somewhat disagree (2) | 5.1 | 6.3 | 11.0
  Strongly disagree (1) | 6.3 | 3.8 | 7.3
  No opinion | 2.5 | 1.3 | 2.4

25. Secondary Outcome: My Eye Appears Healthy - 2 Minutes After First Application
Description: as for outcome 9
Time Frame: 2 minutes after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 46.8 | 44.3 | 42.7
  Somewhat agree (4) | 40.5 | 34.2 | 37.8
  Neither agree or disagree (3) | 8.9 | 13.9 | 13.4
  Somewhat disagree (2) | 1.3 | 5.1 | 3.7
  Strongly disagree (1) | 0 | 1.3 | 1.2
  No opinion | 2.5 | 1.3 | 1.2

26. Secondary Outcome: My Eye Appears Healthy - 10 Hours After First Application
Description: as for outcome 9
Time Frame: 10 hours after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 48.1 | 50.6 | 48.8
  Somewhat agree (4) | 29.1 | 27.8 | 28.0
  Neither agree or disagree (3) | 11.4 | 12.7 | 13.4
  Somewhat disagree (2) | 5.1 | 6.3 | 6.1
  Strongly disagree (1) | 0 | 0 | 1.2
  No opinion | 5.1 | 2.5 | 2.4

27. Secondary Outcome: My Eye Appears Healthy - 12 Hours After First Application
Description: as for outcome 9
Time Frame: 12 hours after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 54.4 | 51.9 | 47.6
  Somewhat agree (4) | 29.1 | 22.8 | 28.0
  Neither agree or disagree (3) | 11.4 | 11.4 | 18.3
  Somewhat disagree (2) | 1.3 | 5.1 | 2.4
  Strongly disagree (1) | 0 | 1.3 | 0
  No opinion | 2.5 | 5.1 | 2.4

28. Secondary Outcome: My Eye Feels Cool - 2 Minutes After First Application
Description: as for outcome 9
Time Frame: 2 minutes after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 29.1 | 20.3 | 29.3
  Somewhat agree (4) | 40.5 | 44.3 | 32.9
  Neither agree or disagree (3) | 24.1 | 24.1 | 25.6
  Somewhat disagree (2) | 6.3 | 7.6 | 8.5
  Strongly disagree (1) | 0 | 2.5 | 2.4
  No opinion | 0 | 1.3 | 1.2

29. Secondary Outcome: My Eye Feels Cool - 10 Hours After First Application
Description: as for outcome 9
Time Frame: 10 hours after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 24.1 | 20.3 | 13.4
  Somewhat agree (4) | 29.1 | 36.7 | 34.1
  Neither agree or disagree (3) | 21.5 | 25.3 | 23.2
  Somewhat disagree (2) | 17.7 | 10.1 | 14.6
  Strongly disagree (1) | 2.5 | 6.3 | 13.4
  No opinion | 2.5 | 1.3 | 1.2

30. Secondary Outcome: My Eye Feels Cool - 12 Hours After First Application
Description: as for outcome 9
Time Frame: 12 hours after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 20.3 | 22.8 | 17.1
  Somewhat agree (4) | 29.1 | 27.8 | 29.3
  Neither agree or disagree (3) | 31.6 | 30.4 | 24.4
  Somewhat disagree (2) | 12.7 | 10.1 | 17.1
  Strongly disagree (1) | 5.1 | 5.1 | 11.0
  No opinion | 0 | 2.5 | 1.2

31. Secondary Outcome: My Eye Appears to Sparkle - Baseline
Description: as for outcome 9
Time Frame: Baseline
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 3.8 | 6.3 | 9.8
  Somewhat agree (4) | 24.1 | 20.3 | 19.5
  Neither agree or disagree (3) | 34.2 | 38.0 | 35.4
  Somewhat disagree (2) | 11.4 | 8.9 | 7.3
  Strongly disagree (1) | 7.6 | 11.4 | 13.4
  No opinion | 19.0 | 15.2 | 14.6

32. Secondary Outcome: My Eye Appears to Sparkle - 2 Minutes After First Application
Description: as for outcome 9
Time Frame: 2 minutes after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 6.3 | 8.9 | 14.6
  Somewhat agree (4) | 34.2 | 26.6 | 20.7
  Neither agree or disagree (3) | 30.4 | 35.4 | 37.8
  Somewhat disagree (2) | 5.1 | 6.3 | 4.9
  Strongly disagree (1) | 3.8 | 7.6 | 8.5
  No opinion | 20.3 | 15.2 | 13.4

33. Secondary Outcome: My Eye Appears to Sparkle - 10 Hours After First Application
Description: as for outcome 9
Time Frame: 10 hours after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 19.0 | 15.2 | 17.1
  Somewhat agree (4) | 29.1 | 34.2 | 28.0
  Neither agree or disagree (3) | 27.8 | 31.6 | 29.3
  Somewhat disagree (2) | 10.1 | 2.5 | 7.3
  Strongly disagree (1) | 1.3 | 7.6 | 9.8
  No opinion | 11.4 | 8.9 | 8.5

34. Secondary Outcome: My Eye Appears to Sparkle - 12 Hours After First Application
Description: as for outcome 9
Time Frame: 12 hours after first application
Population: Intent-to-treat set
Measure: Number; unit: Percentage of participants
Units Other Than Participants: Eyes
Arm/Group | F# PF004390 Eye Drops | F# 13418-148 Eye Drops | F#13418-158 Eye Drops
Number analyzed (Participants) | 79 | 79 | 82
Number analyzed (Eyes) | 79 | 79 | 82
Percentage of participants
  Strongly agree (5) | 17.7 | 13.9 | 19.5
  Somewhat agree (4) | 29.1 | 25.3 | 24.4
  Neither agree or disagree (3) | 31.6 | 38.0 | 26.8
  Somewhat disagree (2) | 8.9 | 5.1 | 9.8
  Strongly disagree (1) | 2.5 | 7.6 | 11.0
  No opinion | 8.9 | 8.9 | 8.5

ADVERSE EVENTS:
Time Frame: Through 24-hour end-of-study visit; + up to 30 days for unresolved adverse events; +30 days for serious adverse events
Description: AEs were systematically collected during the study. AEs that were unresolved upon completion or termination from the study were followed for up to 30 calendar days until the event or its sequelae resolved or stabilized. Serious AEs were collected through 30 calendar days after the participant's last study visit.
Arm/Group | F#13418-148/F#13418-158 | F#13418-148/F#PF004390 | F#13418-158/F#PF004390
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/38 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/38 | 0/41
Other Adverse Events (participants affected / at risk) | 0/41 | 0/38 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Prior to submission for publication, PI was to provide sponsor with ≥ 60 days for publication review. No publication that included sponsor confidential information was to be submitted without sponsor's prior written consent. If requested, the PI was to withhold publication for up to 60 additional days to allow for patent application filing.

DOCUMENTS (2):
  • Study Protocol (2017-03-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT03198000/Prot_002.pdf
  • Statistical Analysis Plan (2017-06-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT03198000/SAP_003.pdf